CLINICAL TRIAL: NCT06368739
Title: Evaluation of Medicaid Grocery Gift Cards & Nutrition Education Program for Pregnant Women on Maternal and Infant Outcomes
Brief Title: Evaluation of Medicaid Food & Nutrition Support Program for Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Driscoll Health Plan (Unknown)
Responsible Party: Principal Investigator, Maninder Kahlon, Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00005622
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy Related; Financial Gift; Nutrition, Healthy
Keywords: gift card; nutrition education; nutrition consultation; food purchase; recipe; telephone; medicaid; health claims
MeSH Terms: conditions — Gift Giving

STUDY DESIGN:
Intervention Model Description: From the eligible population, DHP randomly selected a subset of approximately 500 women during the pilot period, from which approximately 200 were in the program, the "exposed group." The women who were covered during the same period but were not selected were not exposed to the program and will compose the "comparison group."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurture + regular benefits (exposed group) (Experimental): 1. Monthly packages sent every four weeks until end of pregnancy with maximum of eight packages. Each package includes:
     US $40 grocery store gift card A healthy eating information sheet selected from Brighter Bites project. (https://brighterbites.org/).
     A set of three recipes. Nutrition-related Frequently Asked Questions (in four of eight packages).
  2. Two 30-minute telephonic nutritional consultations. Designed by a Registered Dietitian Nutritionist (RDN) who trained a bilingual nutrition specialist to deliver the consultations. Topics revolved around healthy eating during pregnancy, such as food choices, portion sizes, budget-friendly shopping, food safety, and food preparation. No nutrition therapy advice to manage diseases was provided.
  3. Regular benefits Includes regular healthcare services offered as part of the health plan coverage with Medicaid/CHIP.
  Interventions: Behavioral: Nurture program; Other: Regular benefits
- Regular benefits (comparison group) (Active Comparator): Regular benefits
  Includes regular healthcare services offered as part of the health plan coverage with Medicaid/CHIP.
  Interventions: Other: Regular benefits

INTERVENTIONS:
Behavioral: Nurture program — 1. Nurture Monthly Packages: Sent every four weeks until the member reaches the end of pregnancy (delivery or other reasons, e.g., miscarriage), with a maximum of eight packages. Each package includes:
     * A US$40 gift card (2 x $20 each) to a grocery store.
     * A healthy eating information sheet selected from Brighter Bites project (https://brighterbites.org/).
     * A set of three recipes.
     * Nutrition-related Frequently Asked Questions (included in four out of the eight packages).
  2. Two 30-Minute Nutritional Consultations over the phone: Designed by a Registered Dietitian Nutritionist (RDN) who trained a bilingual nutrition specialist to deliver the consultations. Topics revolved around healthy eating during pregnancy, such as food choices, portion sizes, budget-friendly shopping, food safety, and food preparation. No nutrition therapy advice to manage diseases was provided.
  Arms: Nurture + regular benefits (exposed group)
Other: Regular benefits — Includes regular healthcare services offered as part of the health plan coverage with Medicaid/CHIP.

SUMMARY:
With funding from the Episcopal Health Foundation, the researchers will conduct a secondary data analysis to evaluate the impact of Driscoll Health Plan's Nurture program for pregnant members using claims data.

DETAILED DESCRIPTION:
This record describes a quality improvement program (called "Nurture") piloted by Driscoll Health Plan, which included nutrition education and food purchase support offered to a subset of pregnant women aged 30 years and above and covered by the Medicaid Managed Care Organization (MCO) plan in their "STAR" and "CHIP" programs during October 2022 and July 2023.

Factor Health lab at Dell Medical School at the University of Texas at Austin will do a secondary data analysis to evaluate the impact of DHP's program.

Driscoll Health Plan (DHP) is a non-profit, community-based health insurance plan that provides coverage to South Texas and the Rio Grande Valley communities. Their insurance products include STAR Medicaid, STAR Kids, CHIP, and CHIP Perinatal.

With input from Factor Health lab at Dell Medical School, DHP introduced the Nurture program for its members as a quality improvement initiative, designed to expand members' access to nutrition education and food purchase support to improve health and pregnancy outcomes.

Nurture included up to 8 packages mailed every four weeks until the member reaches the end of pregnancy. Each package included USD $40 in the form of gift cards to a large-chain grocery store, a healthy eating information sheet selected from Brighter Bites (https://brighterbites.org/), a set of three recipes, and nutrition-related Frequently Asked Questions during pregnancy (in four out of the eight packages). Members also received two 30-minute nutritional consultations over the phone.

Members had the flexibility to opt out of the program at any time and discontinue receiving packages. Consultations were optional. If they opted out, they continued to receive the DHP benefits as part of their regular coverage.

ELIGIBILITY:
Inclusion Criteria:

* Member of Driscoll Health Plan
* Pregnant
* Aged 30 or older

Exclusion Criteria:

* Not a member of Driscoll Health Plan
* Not pregnant
* Younger than 30 years of age

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Composite outcome 1: Adverse health events during pregnancy | At pregnancy delivery
  Composite includes health claims (paid or non-paid) with codes related to:
  * Gestational Diabetes Mellitus
  * Excessive weight gain during pregnancy
  * Pregnancy-associated hypertension
Composite outcome 2: Adverse health events at birth and newborn-related | At pregnancy delivery
  Composite includes health claims (paid or non-paid) with codes related to:
  * Pre-term birth (<37 weeks)
  * Neonatal Intensive Care Unit (NICU)
  * Small for gestational age
  * Large for gestational age
  * Stillbirths

OTHER OUTCOMES:
Emergency Department visits | At pregnancy delivery
  Health claims with codes related to visits to emergency department.
Cost (outpatient) | At pregnancy delivery
  Cost of outpatient services (e.g., primary care visits, screening) as available in paid health claims.
Cost (inpatient) | At pregnancy delivery
  Cost of inpatient services (e.g., delivery) as available in paid health claims.
Cost (pharmacy/medication) | At pregnancy delivery
  Cost of medication as available in paid health claims.
Cost (total) | At pregnancy delivery
  Total cost of care as available in paid health claims.
Delivery mode (vaginal, C-section) | At pregnancy delivery
  Health claims with codes related to mode of delivery.
Birthweight | At pregnancy delivery
  Requested from hospital's electronic health records (as available)
Prenatal visits | At pregnancy delivery
  Number of prenatal visits during study pregnancy
Gift card usage | 30 days after inactive from program
  Binary response was gift card fully used
Nutritional consults attended | At pregnancy delivery
  Categorical description of nutritional consults attended, both/one/none

CONTACTS AND LOCATIONS:
Locations (1):
- Driscoll Health Plan, Corpus Christi, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No data will be shared with other researchers.

REFERENCES:
- See also: Source of nutrition education materials included in the Nurture packages mailed to participants. — https://brighterbites.org/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT06368739/Prot_SAP_000.pdf